CLINICAL TRIAL: NCT04008784
Title: Improvement of Short Term Outcome of Mild to Moderate Atopic Dermatitis Using a Combination Treatment of Crisaborole Ointment, 2% and a Concomitant Topical Corticosteroid Over a 8 Week Period
Brief Title: Improvement of Short Term Outcome of Mild to Moderate Atopic Dermatitis Using a Combination of Crisaborole and a Concomitant Topical Corticosteroid Over a 8 Week Period
Status: Completed | Type: Observational
Sponsor: Clinical Research Center of the Carolinas (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CRCC-2019-001
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole; Triamcinolone Acetonide; Ointments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Crisaborole 2% Topical Application Ointment [EUCRISA]: Crisaborole 2% Topical Application Ointment [EUCRISA] applied twice a day for 8 weeks
  Interventions: Drug: Crisaborole 2% Topical Application Ointment [EUCRISA]
- Crisaborole 2% plus Triamcinolone Acetonide 0.1%Ointment: Crisaborole 2% plus Triamcinolone Acetonide 0.1% Ointment applied twice a day for the first 2 weeks, followed by Crisaborole 2% alone applied twice a day for the following 6 weeks
  Interventions: Drug: Crisaborole 2% Topical Application Ointment [EUCRISA]; Drug: Triamcinolone Acetonide 0.1% Ointment

INTERVENTIONS:
Drug: Crisaborole 2% Topical Application Ointment [EUCRISA] — Ointment
Drug: Triamcinolone Acetonide 0.1% Ointment — Topical Corticosteroid
  Groups: Crisaborole 2% plus Triamcinolone Acetonide 0.1%Ointment

SUMMARY:
This trial is a single-center two arm, open label observational prospective study, that will evaluate the safety and efficacy of crisaborole ointment, 2% alone compared to a combination therapy of crisaborole and a topical corticosteroid (Triamcinolone Acetonide Ointment, 0.1%) over a 8 week period for the treatment of mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
Male and female subjects, ages 2 to 79 with mild to moderate atopic dermatitis and having an Investigator's Global Assessment Score on a five point scale of 2 or 3 will be enrolled.

Sixteen subjects will be enrolled and randomized 1:1. Eight subjects will be randomized to receive crisaborole alone which will be applied twice daily, once in the morning and once in the evening for 8 weeks. Eight subjects will be randomized to receive a combination therapy of a topical corticosteroid (Triamcinolone Acetonide Ointment, 0.1% and crisaborole ointment, 2% which will be applied twice a day, once in the morning and once in the evening for the first two weeks, followed by crisaborole alone for the following six weeks.

Subjects who meet the inclusion criteria and none of the exclusion criteria at the Screening visit will return to the clinic on Week 0 for Baseline measures and to start treatment which will continue for a period of 8 weeks. Subjects who do not need to undergo a wash-out period may combine the Screening visit and Baseline visit.

Screened subjects requiring a wash-out period (up to 4 weeks) prior to baseline measurements and beginning treatment will attend a total of 4 visits.

Following the Baseline (Week 0) visit, all subjects will report to the clinic for efficacy and safety evaluations at weeks 2, 4 and at the end of study at week 8.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 2 to 79 years of age with confirmed diagnosis of atopic dermatitis
* Clinical diagnosis of atopic dermatitis that has been clinically stable for ≥1 month
* Total body surface area (BSA) of atopic dermatitis involvement ≤35%, excluding involvement of the scalp.
* Patient or patient's parent(s)/legal representative guardian must be willing and able to apply study medications as directed, comply with study instructions, and commit to attending all visits.
* Females of childbearing potential must use at least one highly effective method of birth control. Males with partners of childbearing potential should inform them of their participation in this clinical study and use highly effective methods of birth control during the study.
* Patient or patient's parent(s)/legal representative must be capable of giving written informed consent or verbal assent, as applicable, which includes compliance with the requirements and restrictions listed in the consent/assent form; written informed consent must be obtained prior to any study related procedures.

Exclusion Criteria:

* Concurrent or recent use of certain topical or systemic medications or phototherapy without a sufficient washout period.
* Active or potentially recurrent dermatologic condition other than atopic dermatitis in the target lesion area that may confound evaluation.
* Significant confounding conditions as assessed by study doctor.
* History or evidence of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* Participated in any other trial of an investigational drug or device within 30 days or participation in a research study concurrent with this study
* Pregnancy or lactation.
* History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or medical monitor, contraindicates their participation.
* Patients with active infection in atopic dermatitis areas requiring antibiotics, antifungals, or antiviral agents within 7 days of Baseline (Day 0).
* Patients with pruritus due to conditions other than atopic dermatitis that, in the opinion of the Investigator, would either interfere with study evaluations or affect the safety of the patient.
* History of and/or concurrent condition of serious hypersensitivity (anaphylactic shock or anaphylactoid reaction) to PDE4 inhibitors.
* Use of any prohibited medication. Prohibited concomitant medications, therapy, etc.

during the defined period are as listed below. If a patient requires any of these medications throughout the study period, he/she may be excluded from or discontinued from the study, at the discretion of the Investigator and medical monitor. • From 6 Months prior to the first application of the study drug: Biological products that might have significantly affected the evaluation of atopic dermatitis condition (e.g., tumor necrosis factor [TNF] inhibitors, antiimmunoglobulin [Ig]E antibodies, anti-CD20 antibodies, anti-interleukin [IL]-4 receptor

• From 21 days prior to the first application of study drug: Corticosteroid preparations (oral, injection, and suppository preparations) and topical corticosteroids that were classified as super-high potency (clobetasol propionate).

Oral preparations and injections of immunosuppressants (cyclosporine, methotrexate, azathioprine, tacrolimus, etc.); Excessive sun exposure, tanning booth, other ultraviolet (UV) light source and phototherapy including psoralen and ultraviolet A (PUVA) therapy. • From 14 days prior to the first application of the study drug: any other topical phosphodiesterase 4 (PDE4) inhibitor; Tacrolimus and pimecrolimus cream and/or ointment; Topical corticosteroids that were classified as low, medium, or high potency (e.g., fluocinonide, triamcinolone acetonide, desonide, hydrocortisone).

Eye drops and nasal preparations are allowed.

• From 7 days prior to the first application of the study drug: Oral or intravenous antibiotics, antifungal or antivirus medications Antihistamines/anti-allergics (oral, topical and injections): diphenhydramine, chlorpheniramine maleate, hydroxyzine).

* Visible skin disease or damaged skin at the application site
* Psoriasis and/or active atopic dermatitis/eczema
* Not willing to refrain from using any topical/systemic analgesics such as aspirin
* Pregnant, plan to become pregnant during the study, or are breast-feeding a child
* Using medication which, in the opinion of the investigative personnel, will interfere with the study results, including anti-inflammatory medications
* Any known sensitivity to adhesives;
* Received treatment for any type of internal cancer within 5 years prior to study entry; or have a history of, or are currently being treated for skin cancer;
* Has unstable AD or any consistent requirement for high-potency topical corticosteroids to manage AD signs and symptoms
* Has any clinically significant medical disorder, condition, or disease or clinically significant physical examination finding at Screening that may interfere with study objectives/safety of participants

Ages: 2 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients age 2 to 79 years of age with confirmed diagnosis of atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | Week 8
  2 grade or greater improvement from baseline

SECONDARY OUTCOMES:
Improvement in Patient Itching | Week 8
  Visual Analog Scale (1-10) for Itching improvement

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schlesinger, MD, Principal Investigator — Clinical Research Center of the Carolinas
Locations (1):
- Clinical Research Center of the Carolinas, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weidinger S, Novak N. Atopic dermatitis. Lancet. 2016 Mar 12;387(10023):1109-1122. doi: 10.1016/S0140-6736(15)00149-X. Epub 2015 Sep 13. PMID 26377142
- [Background] Patel NU, Felix K, Reimer D, Feldman SR. Calcipotriene/betamethasone dipropionate for the treatment of psoriasis vulgaris: an evidence-based review. Clin Cosmet Investig Dermatol. 2017 Sep 29;10:385-391. doi: 10.2147/CCID.S131727. eCollection 2017. PMID 29033598
- [Background] PL McCormack - American journal of clinical dermatology, 2011 - Springer
- See also: NDA 207695 Risk Assessment Review — http://www.accessdata.fda.gov/drugsatfda_docs/nda/2016/207695Orig1s000RiskR.pdf
- See also: NDA 207695 Clinical Review — http://www.accessdata.fda.gov/drugsatfda_docs/nda/2016/207695Orig1s000MedR.pdf
- See also: Crisaborole FULL PRESCRIPTION INFORMATION — http://www.accessdata.fda.gov/drugsatfda_docs/nda/2016/207695Orig1s000Lbl.pdf